CLINICAL TRIAL: NCT01842893
Title: Randomized, Placebo-controlled Study of Fentanyl ETHYPHARM for Breakthrough Pain in Opioid-treated Patients With Cancer
Brief Title: Efficacy and Safety of Fentanyl ETHYPHARM for Breakthrough Pain in Opioid-treated Patients With Cancer
Acronym: ETHYFYL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethypharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FYL/24019/008
Record Dates: First submitted 2013-04-18; First posted 2013-04-30 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Breakthrough Pain; Cancer
Keywords: fentanyl; breakthrough pain; opioid treated cancer patients
MeSH Terms: conditions — Breakthrough Pain; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl / Placebo (Experimental): After an open-label titration to identify an optimal dose, patients were randomized to 1 of 13 prespecified sequences of 9 tablets (6 fentanyl and 3 placebo)
  Interventions: Drug: Fentanyl Ethypharm

INTERVENTIONS:
Drug: Fentanyl Ethypharm — After an open-label titration to identify an optimal dose, patients were randomized to 1 of 13 prespecified sequences of 9 tablets (6 fentanyl and 3 placebo)

SUMMARY:
The purpose of the study is to assess the clinical effectiveness of Fentanyl ETHYPHARM when used to relieve breakthrough pain (BTP) in opioid-treated cancer patients.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent
2. Malignant solid tumor or a hematological malignancy causing cancer-related pain
3. Background opioid treatment at a stable dose for at least a week
4. One to four episodes of breakthrough pain per day

Main exclusion criteria:

1. Hypersensitivity to fentanyl or to any of the excipients
2. Intrathecal opioids
3. Recent history of substance abuse
4. Recent or planned therapy that would alter pain
5. Moderate or severe hepatic or renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference at 30 minutes (SPID30). | 30 minutes post dose

SECONDARY OUTCOMES:
SPID at 3, 6, 10, 15 and 60 minutes post-dosing | 3, 6, 10, 15 and 60 minutes post-dosing
SPID at 15 and 30 minutes according to the pathophysiology of the pain (neuropathic, nociceptive) | 15 and 30 minutes post dose
Pain Intensity Difference at 3, 6, 10, 15, 30 and 60 minutes after dosing | 3, 6, 10, 15, 30 and 60 minutes after dosing
Pain Relief at 3, 6, 10, 15, 30 and 60 minutes after dosing | 3, 6, 10, 15, 30 and 60 minutes after dosing
The proportion of episodes of BTP that required rescue medication | 15 and 30 minutes post dose
the proportion of episodes with more than 33% and 50% of improvement in Pain Intensity scores | 15 and 30 minutes post dose
Recording of safety data | During all the study duration, an expected average of 8 weeks
  Adverse events, vital signs, urinary pregnancy test

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Care Units, Prague, Czechia

REFERENCES:
- [Derived] Novotna S, Valentova K, Fricova J, Richterova E, Harabisova S, Bullier F, Trinquet F; ETHYFYL Study Group. A randomized, placebo-controlled study of a new sublingual formulation of fentanyl citrate (fentanyl ethypharm) for breakthrough pain in opioid-treated patients with cancer. Clin Ther. 2014 Mar 1;36(3):357-67. doi: 10.1016/j.clinthera.2014.01.006. Epub 2014 Feb 5. PMID 24508417